CLINICAL TRIAL: NCT06779305
Title: Minimally Invasive Procedure Versus Conservative Treatment in the Management of Calcaneal Joint Fractures
Acronym: IMPACT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-PP-14
Record Dates: First submitted 2025-01-10; First posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Calcaneus ; Fracture ; Traumatology
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Minimally invasive surgery group (Experimental)
  Interventions: Procedure: Minimally invasive surgical application of Calcanail®
- Conservative treatment group (Active Comparator)
  Interventions: Procedure: Immobilisation by cast boot

INTERVENTIONS:
Procedure: Minimally invasive surgical application of Calcanail® — The procedure involves making small incisions to insert a specialized nail into the bone to realign and stabilize the fracture. This approach minimizes damage to surrounding tissues, reduces the risk of wound complications, and allows for quicker recovery compared to traditional open surgery. after surgery, the patient will benefit from an immobilisation with a plaster boot without support for 3 weeks, followed by immobilisation with a removable walking boot for 3 weeks with partial support depending on the patient's pain.
  Arms: Minimally invasive surgery group
Procedure: Immobilisation by cast boot — The patient will be immobilised in a plaster cast without support for 3 weeks, followed by immobilisation in a removable walking boot for 3 weeks with partial support depending on the pain.
  Arms: Conservative treatment group

SUMMARY:
Calcaneal fractures, which affect the heel bone, are the most common type of tarsal fractures and often occur in young people, leading to long recovery times and significant social and economic consequences. Traditional treatments include either non-surgical methods, like immobilizing the foot in a cast, or open surgery, which involves a large incision to fix the bone with plates. However, open surgery has a high complication rate, including issues with wound healing. Recent advances have introduced minimally invasive surgical techniques, which use smaller incisions and have shown better results with fewer complications. This study aims to compare two treatment options for displaced calcaneal fractures: a minimally invasive surgery group and a non-surgical treatment group using a plaster boot. The goal is to determine whether minimally invasive surgery provides better outcomes for patients, such as faster recovery, fewer complications, and improved long-term function, to guide future treatment practices. Thus, this is a prospective, randomised comparative study of the management of articular fractures of the calcaneus: conservative treatment versus minimally invasive surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patient aged 18 or over
2. Patient with a posterior articular fracture of the calcaneus Sanders II to IV, less than 15 days old
3. Patient affiliated to a social security scheme,
4. Patient having given written consent following written and oral information.

Exclusion Criteria:

1. Patient with open calcaneal fracture
2. Patient with bilateral calcaneal fracture
3. Patient with extreme varus or valgus impingement of the fibula
4. Patient with associated talar, tibial, femoral and/or pelvic fracture or associated spinal cord injury.
5. Patient unsuitable for loco-regional anaesthesia (LRA).
6. Patient with neuro-psychiatric disorders resulting in an inability to follow a post-surgical or post-immobilisation rehabilitation protocol.
7. Pregnant women
8. Patient protected by law under guardianship or curatorship, or unable to participate in a clinical study under article L. 1121-16 of the French Public Health Code.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-01-16 (Estimated); Primary Completion 2028-01-16 (Estimated); Study Completion 2028-01-16 (Estimated)

PRIMARY OUTCOMES:
To show a significant difference in favour of minimally invasive surgical treatment compared with orthopaedic treatment for displaced articular fractures of the calcaneus. | 1 year follow-up
  The primary endpoint is the American Orthopaedic Foot & Ankle Society (AOFAS) clinical score

SECONDARY OUTCOMES:
Demonstrate the superiority of minimally invasive surgical treatment over orthopaedic treatment on :A reduction in the rate of early complications (skin problems, infections, complex regional pain syndrome) | 1 year follow-up
  The superiority of minimally invasive surgery over orthopaedic surgery in terms of early complications will be assessed by the rate of scar disunions, skin necrosis, complex regional pain syndrome (CRPS) and surgical site infections.
Demonstrate the superiority of minimally invasive surgical treatment over orthopaedic treatment on :A reduction in the rate of late complications (rate of arthrodesis revision) | 1 year follow-up
  Assessment of the superiority of minimally invasive surgical treatment over orthopaedic treatment in terms of late complications will be based on the long-term need for revision surgery or subtalar arthrodesis.
Demonstrate the superiority of minimally invasive surgical treatment over orthopaedic treatment on :Improved anatomical relationships (radiological measurements) | 1 year follow-up
  Assessment of the superiority of minimally invasive surgical treatment over orthopaedic treatment in terms of restoration of calcaneal anatomy will be based on radiological measurements: Bohler angle and Meary angle. The Böhler angle is expressed in degrees and correlates with the recovery or otherwise of the calcaneal morphology. The Meary angle is expressed in degrees and correlates with the recovery or otherwise of the axis of the hindfoot.
Demonstrate the superiority of minimally invasive surgical treatment over orthopaedic treatment on : Improved bootability at 1 year. | 1 year follow-up
  Assessment of the superiority of minimally invasive surgical treatment over orthopaedic treatment with respect to footwear will be assessed by being able to fit into: a) all types of footwear, b) some or c) not being able to fit into footwear.
Demonstrate the superiority of minimally invasive surgical treatment over orthopaedic treatment on :A reduction in the time taken to return to work and sport at 1 year. | 1 year follow-up
  Assessment of the superiority of minimally invasive surgical treatment compared to orthopaedic treatment in terms of whether or not the patient can return to work and sport (binary yes or no answer) at follow-up consultations.
Demonstrate the superiority of minimally invasive surgical treatment over orthopaedic treatment on : An improvement in the patient self-assessment score (SAV) at 1 year. | 1 year follow-up
  Assessment of the superiority of minimally invasive surgical treatment compared to orthopaedic treatment in terms of patient self-evaluation score. This will be based on the SAV Simple Ankle Value (PROMS) score (Appendix II). The assessment question will be "What percentage would you rate the function of your ankle today, if 100% was a normal ankle?". The answer will be on a scale from 0% to 100%, where 100% is normal function.